CLINICAL TRIAL: NCT03422887
Title: Flurbiprofen Axetil and Nalbuphine for Postoperative Pain and Discomfort After Oculoplastic Surgery
Brief Title: Nalbuphine and Flurbiprofen for Oculoplastic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huijing Ye, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201802
Record Dates: First submitted 2018-01-18; First posted 2018-02-06 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Surgery; Anesthesia; Pain
Keywords: postoperative pain; general anesthesia; postoperative discomfort
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Nalbuphine; flurbiprofen axetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- flurbiprofen axetil (Active Comparator): flurbiprofen axetil intraoperative administration 100mg
  Interventions: Drug: Flurbiprofen Axetil
- nalbuphine (Experimental): nalbuphine intraoperative administration 0.1mg/kg
  Interventions: Drug: Nalbuphine
- nalbuphine and flurbiprofen axetil (Experimental): flurbiprofen axetil intraoperative administration 100mg and nalbuphine intraoperative administration 0.1mg/kg
  Interventions: Drug: Nalbuphine and Flurbiprofen Axetil

INTERVENTIONS:
Drug: Nalbuphine — Nalbuphine administration during surgery
  Arms: nalbuphine
Drug: Flurbiprofen Axetil — Flurbiprofen axetil administration during surgery
  Arms: flurbiprofen axetil
Drug: Nalbuphine and Flurbiprofen Axetil — Nalbuphine and Flurbiprofen Axetil administration during surgery
  Arms: nalbuphine and flurbiprofen axetil

SUMMARY:
The purpose of this study is to evaluate the postoperative pain and discomfort using flurbiprofen axetil or nalbuphine administration after oculoplastic surgery under general anesthesia.

DETAILED DESCRIPTION:
In this randomized controlled clinical trial, we evaluated the postoperative analgesic efficacy and adverse effects of flurbiprofen axetil combined with nalbuphine in patients undergoing oculoplastic surgery compared with a single dose of flurbiprofen axetil or nalbuphine.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing oculoplastic surgery
* age between 16 and 75 years
* American Society of Anesthesiologists (ASA) physical status of I-II

Exclusion Criteria:

* serious coexisting disease
* body mass index (BMI) <18.5 or >35
* contraindications or previous adverse reactions to any of the drugs used
* females with a positive pregnancy test
* patients unable to cooperate

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pain 24 hours after recovery | 24 hours after recovery
  Pain levels measured using Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents no pain and 10 represents the worst pain imaginable ; this scale has been confirmed to be sensitive and reliable.Clinically significant postoperative pain was considered serious pain (NRS score ≥5).

SECONDARY OUTCOMES:
Discomfort 24 hours after recovery | 24 hour after recovery
  Discomfort levels were measured using Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents no discomfort and 10 represents the worst discomfort; this scale has been confirmed to be sensitive and reliable. Discomfort was defined as "sensation other than pain" and included nausea, vomiting, headache, and dizziness. Clinically significant postoperative discomfort was considered serious discomfort (NRS score ≥5) any time postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Ye, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided